CLINICAL TRIAL: NCT01306760
Title: The Use of Ketamine as an Anaesthetic During Electroconvulsive Therapy (ECT) for Depression: Does it Improve Treatment Outcome?
Brief Title: The Use of Ketamine as an Anaesthetic During Electroconvulsive Therapy
Acronym: KANECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSO ETM/6
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Depression
Keywords: depression; electroconvulsive therapy; ketamine
MeSH Terms: conditions — Depression | interventions — Ketamine; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): Ketamine used as the anaesthetic during ECT.
  Interventions: Drug: Ketamine
- Propofol (Active Comparator): Propofol, the standard anaesthetic, used during ECT.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ketamine — Ketamine used as the anaesthetic during ECT.
  Other Names: Ketalar
  Arms: Ketamine
Drug: Propofol — The standard anaesthetic used for ECT.
  Other Names: Diprivan 1%
  Arms: Propofol

SUMMARY:
The main aim of this research is to ascertain whether Ketamine would be a more effective anaesthetic for Electroconvulsive Therapy (ECT) than the standard anaesthetic. In doing so the investigators aim to examine the effect of ketamine on ratings of depressive symptoms, the number of required ECT treatments, and the effect of this anaesthetic on memory.

DETAILED DESCRIPTION:
According to WHO statistics, depression is amongst the leading causes of disability worldwide. In its more severe forms, it can be life threatening. The most severe forms of depression, or those that fail to respond to chemical treatment are treated with electroconvulsive therapy (ECT). The treatment is highly effective, and undoubtedly saves lives, but a range of factors, including side effect profile, the necessity for extended hospital care, and stigma, restricts its use.

A recent study has shown that patients who receive ketamine as the anaesthetic for ECT experience an earlier reduction in depressive symptoms and have a greater reduction in depressive symptoms than those receiving propofol (Okamoto et al., 2009). However, in this study eight ECT treatments were given to all participants so it is unknown whether ketamine could have reduced the number of treatments required. Overall, these studies suggest that as well as being a neuroprotective agent; ketamine may also have an antidepressant effect. Given these findings it is hypothesized that the use of ketamine in ECT treatment may reduce the number of ECT sessions required due to this drug's effects on depression ratings.

Our main research question is whether the use of ketamine as the anaesthetic for ECT treatment for depression improves the treatment outcome with respect to speed of response and reduction in side effects when compared to conventional anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 65 years old
* diagnosed with depression and being referred for ECT
* American Society of Anesthesiologists (ASA) score of 1 or 2
* patient receiving ECT on an informal basis (i.e. consenting to treatment and able to give informed consent)

Exclusion Criteria:

* pre-existing neurological disease or cognitive impairment
* co-morbid psychiatric diagnoses
* pre-existing hypertension
* severe respiratory tract disease
* major cardiovascular disease
* pacemakers
* cerebrovascular disorder or malformation
* intracranial mass lesions
* seizure disorder
* intracranial electrode or clips
* intra-ocular pathology
* endocrine or metabolic disease
* severe hematologic disease
* severe fracture
* not able to give consent
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms | After 4th treatment
  The primary outcome measure will be change in depressive symptoms after the fourth ECT treatment. This will be assessed by the change in MADRS and 17-item HDRS scores between start of treatment and this timepoint.

SECONDARY OUTCOMES:
Cognitive side-effects | 2 months
  This will be assessed using the spatial recognition test from the CANTAB battery. This test was chosen as previous research has shown that this test is most sensitive to anterograde memory impairments associated with ECT. By administering this test before, during (after 4th treatment) and after treatment (immediately following and at 1 month follow-up) we will be able to determine whether ketamine can reduce the anterograde memory dysfunction as compared to propofol.
Change in depressive symptoms after treatment | 2 months
  The secondary measure of treatment efficacy will be assessed by the change in MADRS and 17-item HADRS scores immediately after treatment and at 1 month follow-up. Secondly, this will be assessed by the number of treatments required to achieve remission of symptoms, as judged by treating clinicians. By monitoring the number of treatments required we will be able to assess whether ketamine can reduce the number of ECT treatments required.

CONTACTS AND LOCATIONS:
Overall Officials: Ian C Reid, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- Royal Cornhill Hospital, NHS Grampian, Aberdeen, United Kingdom

REFERENCES:
- [Derived] Fernie G, Currie J, Perrin JS, Stewart CA, Anderson V, Bennett DM, Hay S, Reid IC. Ketamine as the anaesthetic for electroconvulsive therapy: the KANECT randomised controlled trial. Br J Psychiatry. 2017 Jun;210(6):422-428. doi: 10.1192/bjp.bp.116.189134. Epub 2017 Mar 2. PMID 28254962